CLINICAL TRIAL: NCT00467467
Title: Alfuzosin Hydrochloride to Relieve Ureteral Stent Discomfort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 0512M78807
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Ureteral Stent Discomfort
MeSH Terms: interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alfuzosin Hydrochloride

SUMMARY:
To assess the impact of alfuzosin vs. placebo on ureteral stent discomfort, urinary symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Undergoing unilateral retrograde ureteroscopy with ureteral stent placement

Exclusion Criteria:

* Significant ureteral trauma
* Concomitant ESWL or other secondary surgical procedure than may impact patient comfort
* Subject with know hypersensitivity to alfuzosin hydrochloride or any component of alfuzosin hydrochloride tablets.
* Pregnancy, nursing mother, or woman of child-bearing age unwilling to take contraception for the duration of the study
* Undergoing bilateral ureteral stenting
* Undergoing antegrade ureteral stenting
* Undergoing simultaneous extracorporeal shockwave lithotripsy
* Urinary infection (fever >101, positive urine culture, many bacteria on urinalysis)
* Primary bladder dysfunction that would impact ability to void without a catheter
* Neurologic dysfunction that would impair pain sensation
* History of chronic pain or substance abuse
* Potent CYP3A4 inhibitors such as ketoconazole, itraconazole, and ritonavir, since alfuzosin blood levels are increased
* Other alpha-blockers
* Phosphodiesterase type 5 inhibitors for erectile function Any subject for whom the principal investigator feels it would not be in his or her best interest to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
effect of study medication on urinary symptoms and quality of life
usage of analgesics/narcotics

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Monga, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States